CLINICAL TRIAL: NCT00259428
Title: EURopean Trial In Atrial Fibrillation or Flutter Patients Receiving Dronedarone for the maIntenance of Sinus Rhythm (EURIDIS)
Brief Title: EURopean Trial In Atrial Fibrillation(AF) or Flutter (AFL) Patients Receiving Dronedarone for the maIntenance of Sinus Rhythm (EURIDIS)
Acronym: EURIDIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD study director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC3153; SR33589B
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Arrhythmia; Anti-Arrhythmia agents
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone 400mg bid (Experimental): dronedarone 400mg tablets
  Interventions: Drug: Dronedarone (SR33589)
- Placebo (Placebo Comparator): matching placebo tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dronedarone (SR33589) — oral administration
  Other Names: Multaq®
  Arms: Dronedarone 400mg bid
Drug: placebo — oral administration
  Arms: Placebo

SUMMARY:
To assess the efficacy of dronedarone versus placebo for the maintenance of normal sinus rhythm after electrical, pharmacological or spontaneous conversion of atrial fibrillation/atrial flutter (AF/AFL).

To assess the efficacy of dronedarone versus placebo on AF/AFL-related symptoms.

To assess the efficacy of dronedarone versus placebo on ventricular rate control in case of AF/AFL recurrence.

DETAILED DESCRIPTION:
This is a double-blind, parallel arm, placebo-controlled, multicentre, multinational, phase III study.

To be eligible, patients must be in normal sinus rhythm at randomisation and must have an ECG-documented history of recent AF/AFL reverted to normal sinus rhythm by electrical, pharmacological or spontaneous conversion

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 21 years or more, in sinus rhythm for at least 1 hour at the time of randomization and with at least one ECG-documented AF/AFL episode in the last 3 months.

Exclusion Criteria:

* MAIN CRITERIA (non-exhaustive list, see protocol for details):

Women of childbearing potential without adequate birth control, Pregnant women, Breastfeeding women, Congestive heart failure NYHA class III or IV, Conditions which increase the risk of severe antiarrhythmic drug side effects, Severe associated conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2001-11; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the time from randomisation to first documented AF/AFL recurrence

SECONDARY OUTCOMES:
- AF/AFL related symptoms collected at the time of ECG/TTEM recording,
- mean ventricular rate during AF/AFL at first recorded AF/AFL recurrence (12-lead ECG or TTEM)
- time from presumed study drug near steady state defined as D5 midnight to first documented AF/AFL recurrence as indicated by ECG/TTEM recording.

CONTACTS AND LOCATIONS:
Overall Officials: ICD Clinical study director (CSD), Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi- Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Result] Singh BN, Connolly SJ, Crijns HJ, Roy D, Kowey PR, Capucci A, Radzik D, Aliot EM, Hohnloser SH; EURIDIS and ADONIS Investigators. Dronedarone for maintenance of sinus rhythm in atrial fibrillation or flutter. N Engl J Med. 2007 Sep 6;357(10):987-99. doi: 10.1056/NEJMoa054686. PMID 17804843
- [Derived] Handelsman Y, Bunch TJ, Rodbard HW, Steinberg BA, Thind M, Bigot G, Konigsberg L, Wieloch M, Kowey PR. Impact of dronedarone on patients with atrial fibrillation and diabetes: A sub-analysis of the ATHENA and EURIDIS/ADONIS studies. J Diabetes Complications. 2022 Jul;36(7):108227. doi: 10.1016/j.jdiacomp.2022.108227. Epub 2022 Jun 8. PMID 35717354